CLINICAL TRIAL: NCT03941990
Title: Impact of 50% Nitrous Oxide Inhalation on Pain Induced by Lumbar Puncture in Emergency: a Double-blind Randomized Controlled Trial.
Brief Title: Lumbar Puncture in Emergency Under Nitrous OXide
Acronym: LENOX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RBHP 2018 MOISSET; 2018-001296-20 (EudraCT Number)
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-05

CONDITIONS: Pain; Anxiety
Keywords: Spinal puncture; Nitrous oxide; Pain; Anxiety; Emergency
MeSH Terms: conditions — Pain; Anxiety Disorders; Emergencies | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to receive experimental treatment (50% N2O - 50% O2) or placebo (Medical Air: 22% O2 - 78% N2).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: double blinding, gas bottles are in undistinguishable boxes, and each gas mask will be filled with odorous ink masking the sweet flavour of N2O. Neither the patient nor the person doing the LP and/or the evaluation of pain and anxiety will know the treatment used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrous oxyde (Experimental): will inhale experimental treatment throughout the entire procedure (50% N2O - 50% 02)
  Interventions: Drug: Fixed 50:50 mixture of nitrous oxide and oxygen
- Placebo (Placebo Comparator): will inhale medical air throughout the entire procedure (22% O2 + N2 Q.S.)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fixed 50:50 mixture of nitrous oxide and oxygen — Gaz inhalation will start 5 minutes before the puncture and will be continued until the end of the procedure.
  Arms: Nitrous oxyde
Other: Placebo — inhale medical air (22% O2 - 78% N2)
  Arms: Placebo

SUMMARY:
Lumbar puncture (LP) is a frequent exam that can cause pain and anxiety. In a scheduled setting, it has been shown that nitrous oxide use during the procedure was able to reduce both pain and anxiety. The goal of this trial is to confirm these results in a more heterogeneous group of patients having a LP, in an emergency setting.

DETAILED DESCRIPTION:
Nitrous oxide (N2O) has analgesic and anxiolytic properties that are known for more than a century. Nonetheless, it's use during lumbar puncture in adults has only been investigated in a scheduled setting.Thus, this study is designed to evaluate the analgesic effect of N2O on the pain induced during lumbar puncture.

Patients with urgent lumbar puncture realized for diagnosis purposes will be randomized in 2 groups. One group will inhale N2O for the 5 minutes before the puncture and during the rest of the procedure. The second group will inhale compressed air during the same period. Neither the investigator realizing the lumbar puncture, nor the patient will know which type of gaz they are inhaling (double-blinding).

The maximal pain level that occurred during the procedure will be evaluated on a Numerical Rating Scale (NRS). NRS will also be used to evaluate the maximal anxiety induced by the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients coming in emergency service who need a lumbar puncture in emergency for a diagnostic purpose
* at least 18
* affiliated to the French state healthcare insurance system
* able to give consent to participation

Exclusion Criteria:

* Previous use of nitrous oxide (medical or recreational)
* Contra-indication to nitrous oxide use
* Face mask phobia
* Stage II obesity (BMI > 35)
* Hemodynamic instability and/or any case when coagulation results cannot be waited
* Cognitive condition defined by a previous Mini Mental State Examination < 24/30
* Confusion or any consciousness disorder that might interfere with judgment or consent
* Patient unable to communicate verbally
* Patient placed under a legal protection measure (tutorship, curatorship or a mandate)
* Any medical condition that might contra-indicate medical research, in physician's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Maximal pain perceived during the lumbar puncture evaluated using a simple numeric 0-10 pain scale | 2-3 minutes after the end of gas inhalation
  Maximal level of pain during lumbar puncture. The patient will be asked to circle the digit that best describes the maximal level of pain felt during the procedure. If the patient is too painful and/or is incapacitated, the collection notebook will be fulfilled by the care provider after asking the following question: "On a scale of 0 to 10, 0 being the absence of pain and 10 the maximal pain you can imagine, what is the digit best describing the maximal pain you felt during the procedure?"

SECONDARY OUTCOMES:
Maximal anxiety perceived during lumbar puncture evaluated using a simple numeric 0-10 scale | 2-3 minutes after the end of gas inhalation
  Proportion of patients with significant anxiety
Side effects | From the beginning of gas inhalation to a minimum of 2 hours later
  Every side effect reported by the patients attributable to gas inhalation during the procedure up to emergency service discharge. Presence, intensity and reversibility will be recorded
Spinal puncture duration | 2-3 minutes after the end of lumbar puncture
  Comparison of LP duration between both groups measured in minutes (from the beginning of gas inhalation to needle removal).
Number of attempts before successful LP | 2-3 minutes after the end of lumbar puncture
  Comparison of number of attempts needed to get spinal fluid, defined as number of needle removals for a single exam.
Patient Satisfaction | 2-3 minutes after the end of gas inhalation
  overall satisfaction based on a 0-10 score and proportion of patients that would accept another lumbar puncture in the same conditions
Blinding quality | 2-3 minutes after the end of gas inhalation
  Assessment of blinding in clinical trials (according to Bang et al. 2004)
Induced cost | through study completion, an average 4 months
  supplementary cost induced by the use of nitrous oxide inhalation for a total of 88 patients throughout the study (gas and consumables such as masks and pipes)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herres J, Chudnofsky CR, Manur R, Damiron K, Deitch K. The use of inhaled nitrous oxide for analgesia in adult ED patients: a pilot study. Am J Emerg Med. 2016 Feb;34(2):269-73. doi: 10.1016/j.ajem.2015.10.038. Epub 2015 Oct 24. PMID 26585197
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Koscielniak-Nielsen Z, Hesselbjerg L, Brushoj J, Jensen MB, Pedersen HS. EMLA patch for spinal puncture. A comparison of EMLA patch with lignocaine infiltration and placebo patch. Anaesthesia. 1998 Dec;53(12):1218-22. doi: 10.1046/j.1365-2044.1998.00608.x. PMID 10193230
- [Background] Lavi R, Yarnitsky D, Rowe JM, Weissman A, Segal D, Avivi I. Standard vs atraumatic Whitacre needle for diagnostic lumbar puncture: a randomized trial. Neurology. 2006 Oct 24;67(8):1492-4. doi: 10.1212/01.wnl.0000240054.40274.8a. PMID 17060584
- [Background] Lukas A, Niederecker T, Gunther I, Mayer B, Nikolaus T. Self- and proxy report for the assessment of pain in patients with and without cognitive impairment: experiences gained in a geriatric hospital. Z Gerontol Geriatr. 2013 Apr;46(3):214-21. doi: 10.1007/s00391-013-0475-y. PMID 23474866
- [Background] Moisset X, Ruet A, Brochet B, Planche V, Jaffeux P, Gilleron V, Ong N, Clavelou P. Who Performs Lumbar Puncture, How Many Do They Perform, How and Why? A Retrospective Study of 6,594 Cases. Eur Neurol. 2016;76(1-2):8-11. doi: 10.1159/000447452. Epub 2016 Jun 24. PMID 27336667
- [Background] Moisset X, Sia MA, Pereira B, Taithe F, Dumont E, Bernard L, Clavelou P. Fixed 50:50 mixture of nitrous oxide and oxygen to reduce lumbar-puncture-induced pain: a randomized controlled trial. Eur J Neurol. 2017 Jan;24(1):46-52. doi: 10.1111/ene.13127. Epub 2016 Sep 25. PMID 27666149